CLINICAL TRIAL: NCT07234474
Title: A Phase I Study of YK012, a Humanized CD19 × CD3 Bispecific Antibody, in Participants With Very High-Risk, Refractory Primary Membranous Nephropathy
Brief Title: A Phase I Study of YK012 in Primary Membranous Nephropathy
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Excyte Biopharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: YK012-3-FDA
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Primary Membranous Nephropathy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ia: YK012 (Experimental): Participants with primary membranous nephropathy will receive ascending doses of YK012 infusion to evaluate the safety and tolerability of YK012, and to determine the Maximum Tolerated Dose (MTD) and Recommended Dose for Expansion (RDE)
  Interventions: Drug: YK012
- Ib: YK012 (Experimental): Participants will receive 2 different doses of YK012 infusion to evaluate the safety and tolerability of YK012 in participants with primary membranous nephropathy and to establish the Recommended Phase II Dose (RP2D).
  Interventions: Drug: YK012

INTERVENTIONS:
Drug: YK012 — YK012 is a bispecific antibody targeting CD19 on B cells and CD3 on T cells leading to T cell-mediated cytotoxicity of malignant B cells

SUMMARY:
The goal of this clinical trial is to evaluate the safety, tolerability, pharmacokinetics(PK), pharmacodynamics (PD), immunogenicity, and preliminary efficacy of YK012 in participants with primary membranous nephropathy (pMN).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 (inclusive), both gender.
* Diagnosed with primary (idiopathic) membranous nephropathy by renal biopsy within 10 years.
* Participants who meet the criteria of very high-risk primary (idiopathic) membranous nephropathy based on 2021 Kidney Disease: Improving Global Outcomes (KDIGO) Clinical Practice Guideline for the Management of Glomerular Diseases and who have failed available therapies for the treatment of pMN.
* eGFR estimated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula is ≥45 mL/min/1.73 m².
* If taking angiotensin-converting enzyme inhibitor (ACEI), angiotensin II receptor blocker (ARB), or Sodium-Glucose Co-Transporter 2 (SGLT-2) inhibitor, the medication dosage must have been stable (≤50% change in dose) for at least 4 weeks prior to screening and continue being stable prior to the initiation of the investigational product.
* Laboratory tests within 7 days prior to enrollment meet the pre-defined criteria.
* Be able to understand and voluntarily participate in this clinical trial with written signed informed consent and available for scheduled visits, treatments, examinations, and other study procedures.

Exclusion Criteria:

* Diagnosed with secondary membranous nephropathy.
* Any prior receipt of protocol-specified pharmacological treatment for membranous nephropathy.
* History of malignant tumor within 5 years prior to screening.
* Poorly controlled hypertension.
* Participants with severe renal insufficiency who have received or require dialysis or kidney transplantation within 6 months prior to the initiation of the investigational product.
* History of diabetic nephropathy confirmed by renal biopsy.
* History of severe or chronic infections within 6 months prior to screening or currently infection requiring systemic antibiotic or antiviral therapy.
* History of cardiovascular event leading to hospitalization within 6 months prior to screening.
* Other severe or poorly controlled diseases that may affect the protocol compliance or efficacy assessments.
* Have active tuberculosis with clear evidence of infection.
* History of substantial organ or bone marrow transplantation.
* Received live vaccination, underwent major surgery, or participated in other clinical trials and applied any other study drugs within 28 days prior to the initiation of the investigational product.
* Hepatitis B surface antigen (HBsAg) positive, or hepatitis B core antibody (HBcAb) positive with hepatitis B virus (HBV) DNA quantification ≥ 1×103 copies/L or ≥ 50 IU/L (HBcAb positive participants require regular HBV DNA testing); Hepatitis C virus (HCV) antibody positive; Human immunodeficiency virus (HIV) seropositive; Syphilis helical antibody positive.
* Peripheral blood CD4+ T-lymphocyte count < 200 cells/μL.
* The peripheral blood B-cell count is below the lower limit of normal.
* Known hypersensitivity to any of the ingredients of YK012.
* Female participants who are pregnant or breastfeeding, or women of childbearing potential (WOCBP) who have a positive pregnancy test result at screening; or those who plan to have children during the trial period and for 12 months after the end of the trial, and those who are unwilling to use one or more physical contraceptive methods during the trial period and for 12 months after the end of the trial.
* Other conditions that the investigator considers inappropriate for participation in this trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2026-10 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Ia: Dose-Limiting Toxicity (DLT) | up to 28 days after the first dose
Adverse Event (AE) | From the first induction to the end of the trial at 53 weeks
Severe Adverse Event | From the first induction to the end of the trial at 53 weeks

SECONDARY OUTCOMES:
Area under the concentration-time curve (AUC0-t) | From 1 hour before the first infusion of YK012 to the end of trial at 53 or 77 weeks
Area under the concentration-time curve from time 0 to ∞ (AUC0-∞) | From 1 hour before the first infusion of YK012 to the end of trial at 53 or 77 weeks
Maximum plasma concentration (Cmax) | From 1 hour before the first infusion of YK012 to the end of trial at 53 or 77 weeks
Time to reach maximum concentration (Tmax) | From 1 hour before the first infusion of YK012 to the end of trial at 53 or 77 weeks
Half-life (t1/2) | From 1 hour before the first infusion of YK012 to the end of trial at 53 or 77 weeks
Apparent clearance (CL) | From 1 hour before the first infusion of YK012 to the end of trial at 53 or 77 weeks
apparent volume of distribution (Vd) | From 1 hour before the first infusion of YK012 to the end of trial at 53 or 77 weeks
Minimum plasma concentration (Cmin) | From 1 hour before the first infusion of YK012 to the end of trial at 53 or 77 weeks
Time to onset and duration of peripheral blood B-cell and B-cell subset depletion | From 1 hour before the first infusion of YK012 to the end of trial at 53 or 77 weeks
Changes in peripheral blood Natural Killer (NK) cells | From 1 hour before the first infusion of YK012 to the end of trial at 53 or 77 weeks
Changes in peripheral blood T cells and T cell subsets (CD4+ T cells, CD8+ T cells) | From 1 hour before the first infusion of YK012 to the end of trial at 53 or 77 weeks
The profile of cytokine changes | From 1 hour before the first infusion of YK012 to the end of trial at 53 or 77 weeks
Positive rates of blood anti-drug antibody (ADA) and neutralizing antibody (Nab) | From 1 hour before the first infusion of YK012 to the end of trial at 53 or 77 weeks
Changes from baseline in 24-hour urine protein during the trial period | From screening to the end of the trial at 53 or 77 weeks
Changes from baseline in estimated glomerular filtration rate (eGFR) during the trial period | From screening to the end of the trial at 53 or 77 weeks
Changes from baseline in anti-phospholipase A2 receptor (PLA2R) antibody titer during the trial period | From screening to the end of the trial at 53 or 77 weeks
Proportion of participants achieving overall renal remission (ORR) | From screening to the end of the trial at 53 or 77 weeks
Proportion of participants achieving Complete Response (CR) and Partial Response (PR) | From screening to the end of the trial at 53 or 77 weeks
Proportion of participants achieving immunological remission | From screening to the end of the trial at 53 or 77 weeks
Time to achieve CR | From screening to the end of the trial at 53 or 77 weeks
Time to achieve ORR | From screening to the end of the trial at 53 or 77 weeks
Duration of CR | From screening to the end of the trial at 53 or 77 weeks
Duration of ORR | From screening to the end of the trial at 53 or 77 weeks
Proportion of participants with treatment failure | From screening to the end of the trial at 53 or 77 weeks
Proportion of participants who relapsed | From screening to the end of the trial at 53 or 77 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Minghui Zhao, Principal Investigator — Peking University First Hospital